CLINICAL TRIAL: NCT03760757
Title: Effectiveness of Two Different Forms of Marine Oil, Derived From the New Zealand Green Lipped Mussel and Krill Oil, on Indirect Markers of Muscle Damage and Soreness During Recovery From Muscle Damaging Exercise in Untrained Men
Brief Title: Effectiveness of Two Different Forms of Marine Oil on Indirect Markers of Muscle Damage and Soreness in Untrained Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tim Mickleborough, Professor, Kinesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1809579862
Record Dates: First submitted 2018-11-07; First posted 2018-11-30 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Inflammation; Muscle
Keywords: krill oil; DOMS; EIMD (exercise induced muscle damage)
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — PCSO-524

STUDY DESIGN:
Intervention Model Description: Randomized controlled non-inferiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCSO-524® (no krill oil) (Experimental): Four total capsules per day (2 in the morning; 2 at night) for 29 days. Amounts per day equal to 800 mg olive oil, 400 mg lipid extract (~58 mg EPA and 44 mg DHA) and 1.8 mg vitamin E (d-alpha-tocopherol).
  Interventions: Dietary Supplement: PCSO-524®
- ESPO-572® (75% PCSO-524®, 25% krill oil) (Experimental): Four total capsules per day (2 in the morning; 2 at night) for 29 days. ESPO-572®, a 75/25% PCSO-24®/Krill oil blend. Each capsule of the ESPO-572® contains green lipped mussel oil, krill oil, olive oil and vitamin E.
  Interventions: Dietary Supplement: ESPO-572®

INTERVENTIONS:
Dietary Supplement: ESPO-572® — ESPO-572® is the same as PCSO-524®, except it has krill oil added to it.
  Arms: ESPO-572® (75% PCSO-524®, 25% krill oil)
Dietary Supplement: PCSO-524® — PCSO-524® (Lyprinol®/Omega XL®) is a nutritional supplement containing a patented extract of highly condensed form of stabilized marine lipids from the New Zealand green lipped mussel (Perna canaliculus) that is combined with olive oil and vitamin E. This marine oil lipid and omega-3 polyunsaturated fatty acid (PUFA) blend is a diverse mixture of sterol esters, sterols, polar lipids, triglycerides, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) (split between the triacylglycerol and polar lipid classes), and free fatty acids.
  Arms: PCSO-524® (no krill oil)

SUMMARY:
To evaluate the effects of PCSO-524®, and a blend of PCSO-24® (75%) and krill oil (25%) (ESPO-572®), on indirect markers of muscle damage, inflammation and soreness during recovery from muscle damaging exercise in untrained men.

DETAILED DESCRIPTION:
The study will be conducted as a randomized, parallel group trial over 29 days. A total of 50 untrained male subjects will participate in this study. Subjects will be classified as 'untrained' if they exercise less than three times per week for less than 30 min during each session. Subjects will be randomly assigned to either a green-lipped mussel oil blend (PCSO-524® supplementation group, n = 25) or a 75/25% PCSO-24®/Krill oil blend group (ESPO-572® supplementation group, n = 25). Supplementation will begin 26 days before an eccentric exercise bout (downhill running, designed to induce muscle damage and continue for 3 days following the muscle damaging exercise bout).

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include males (18 to 30 years), determined to be low risk (as determined by ACSM's Guidelines for Exercise Testing and Prescription (American College of Sports Medicine., Thompson, Gordon, & Pescatello, 2010)
* BMI<30 (not obese) by a modified physical activity readiness questionnaire (PAR-Q),
* Classified as 'untrained' defined by not habitually exercising more than 3x/week. In order to participate subjects would be allowed to exercise not more than three days a week. Each of the exercise sessions must not be longer than 30 minutes and cannot include downhill or uphill running.

Exclusion Criteria:

* History of asthma or exercise-induced asthma, COPD, interstitial lung diseases, or cystic fibrosis, dyspnea
* History of downhill running training or other eccentric endurance exercise within the past 3 months
* History of fish oil or other omega-3 nutritional supplements within the last 3 months
* History of significant pain in hips or knees
* Current participation in a strength training program or having participated in a strength training program within 60 days before the study
* Regular use of anti-inflammatory medication or nutritional supplements (e.g. ketorolac, celecoxib, creatine, protein drinks, amino acids, fish oil or vitamins)
* Current daily use of anti-inflammatory medication such as Tylenol, Advil, or Aleve.
* Allergies to fish, seafood, or shellfish
* Family or personal history of cardiac, peripheral vascular, or cerebrovascular disease.
* A diabetic or experience shortness of breath as determined by the modified PAR_Q.
* In addition to screening subjects for known cardiovascular disease, or signs and symptoms of pulmonary metabolic disease, subjects will be excluded if their values are outside ACSM's guidelines for cardiovascular disease risk as outlined in Figure 2. This would place subjects as low risk. Researchers will be screening based on age, family history of heart attacks, exposure to cigarette smoke, obesity, hypertension, dyslipidemia and pre-diabetes. Since subjects are recruited as sedentary, this a positive risk factor for CVD. Subjects will be screened for dyslipidemia and will be accepted into the study if their values are for low-density lipoprotein (LDL-C) cholesterol less than 130 mg dL-1 (3.37 mmol·L-1) or a total serum cholesterol value of less than 200 mg·dL-1 (5.18mmol L-1) or and HCL-C is greater or equal to 40 mg·dL-1 (1.55mmol L-1). Please note that this will not change the subjects risk status and they will be still classified as low risk. Subjects should not be currently taking and cholesterol lowering medication such as: Atorvastatin (Lipitor), Fluvastatin (Lescol), Lovastatin (Mevacor), Pravastatin (Pravachol), Simvastatin (Zocor), Rosuvastatin (Crestor)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Creatine Kinase | Four days
  Muscle damage markers: Muscle creatine kinase will be measured using a Beckman DU® Spectrophotometer (Beckman Coulter Inc., Brea, CA) at 360nm using a fluorometric assay kit (Cayman Chemicals, Ann Arbor, MI).
  Units: ng/mL
Skeletal muscle slow troponin I | Four days
  Muscle damage markers: Skeletal muscle slow troponin I, (Novus Biologicals LLc., Littleton, CO).
  Units: ng/mL
Interleukin-1 Beta | Four days
  Muscle inflammation markers: Interleukin-1 Beta (Cayman Chemicals, Ann Arbor, MI) will be analyzed using enzyme-linked immunoassay (ELISA).
  Units: pg/mL
Tumor necrosis factor-alpha | Four days
  Muscle inflammation markers: Tumor necrosis factor-alpha (Cayman Chemicals, Ann Arbor, MI) will be analyzed using enzyme-linked immunoassay (ELISA).
  Units: pg/mL
Isometric torque | Four days
  Isometric torque: Isometric torque assessment of the dominant leg extensors will be conducted at a knee angle of 80°flexion (measured by a goniometry) using a Cybex Isokinetic System (Medway, MA).
  Units: Nm
Range of motion | Four days
  Measurement of knee flexion range of motion
  Units: degrees
Swelling | Four days
  Limb girth measurements are used to test for the presence of swelling/edema within a muscle.
  Units: percentage change from baseline
Delayed onset muscle soreness | Four days
  Visual analog scale of muscle soreness (delayed onset muscle soreness; DOMS) - Knee extensor soreness will be assessed using a visual analogue scale with "no soreness" indicated at one end (score 0) and "unbearably painful" at the other (score 10).
  Units: Arbitrary units
Pressure pain threshold | Four days
  A hand-held pressure algometer (Algometer®, Somedic Sales, Hörby, Sweden) will be used to monitor pressure induced pain at five specific sites on the quadriceps.
  Pressure pain threshold units: percentage change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Mickleborough, Ph.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mickleborough TD, Sinex JA, Platt D, Chapman RF, Hirt M. The effects PCSO-524(R), a patented marine oil lipid and omega-3 PUFA blend derived from the New Zealand green lipped mussel (Perna canaliculus), on indirect markers of muscle damage and inflammation after muscle damaging exercise in untrained men: a randomized, placebo controlled trial. J Int Soc Sports Nutr. 2015 Feb 19;12:10. doi: 10.1186/s12970-015-0073-z. eCollection 2015. PMID 25722660